CLINICAL TRIAL: NCT03111472
Title: Development and Evaluation of a Self-management Guide for Community-dwelling People With Parkinson's Disease Who Fall and Their Informal Caregivers
Brief Title: Development and Evaluation of a Guide to Help People With Parkinson's and Their Caregivers to Self-manage Falling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25364
Record Dates: First submitted 2017-03-07; First posted 2017-04-12 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Parkinson Disease; Accidental Fall
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: 30-40 participants will receive the intervention. The intervention will be a guide to help people with Parkinson's and their caregivers to self-manage falls. There will be no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-management guide for falls in Parkinson's (Experimental): A guide for people with Parkinson's and their caregivers to self-manage falls.
  Interventions: Other: Self-management guide for people with Parkinson's who fall and their informal caregivers

INTERVENTIONS:
Other: Self-management guide for people with Parkinson's who fall and their informal caregivers — The self-management guide will be developed utilising information from people with Parkinson's, informal caregivers of people with Parkinson's, healthcare professionals and a systematic review of self-management interventions for people with Parkinson's who fall.

SUMMARY:
This study will investigate whether it is possible, through the development and evaluation of a self-management guide, to improve health related quality of life and concern of falling in people with Parkinson's disease who fall, and reduce caregiver burden in their informal caregivers.

DETAILED DESCRIPTION:
This study will progress through four phases

Phase One

Establish the needs and preferences of people with Parkinson's (PwP) who fall and their informal caregivers for the effective self-management of falls. This will be achieved through questionnaires distributed to 30-40 PwP and their caregivers, with responses analysed through the use of descriptive statistics. A purposive sample of participants, selected through responses to the questionnaire, will be invited to participate in semi-structured interviews. Interviews will be conducted until data saturation has been achieved. These interviews will seek to further identify the thoughts and experiences of PwP and their caregivers in relation to falling, with responses analysed through thematic analysis.

Phase Two

Establish the needs and preferences of PwP who fall and their informal caregivers for the effective self-management of falls, as perceived by healthcare professionals specialising in the care of PwP. This will be achieved through semi-structured interviews and focus groups with 10 healthcare professionals involved in the care of PwP who fall. The interviews will be analysed with thematic analysis.

Phase Three

Development of a prototype of a self-management guide utilising information from phases one and two alongside a systematic review of self-management interventions for people with Parkinson's who fall. The prototype will be distributed to 6-8 dyads of PwP who fall and their caregivers. Feedback will be sought in the form of a questionnaire, with responses analysed through the use of descriptive statistics, and the guide modified accordingly.

Phase Four

Mixed methods acceptability and feasibility study of the modified version of the guide; with a before and after comparison of health related quality of life and concern of falling in PwP, and of caregiver burden in their informal caregivers.

The guide will be distributed to 30-40 pairings of PwP who fall and their caregivers. Baseline assessments of health related quality of life (Parkinson's disease questionnaire 8, PDQ8) and of caregiver burden (Zarit Burden Interview short version) will be completed.

After three months, participants will complete feedback questionnaires to assess the acceptability and the feasibility of the guide, and will repeat the PDQ8 and zarit burden Interview short version . The responses to the questionnaires will be analysed through the use of descriptive statistics, with a before and after comparison of health related quality of life and of caregiver burden.

A purposive sample of participants, selected through their responses to the questionnaires, will be invited to participate in semi-structured interviews, to further explore their thoughts about the guide. Interviews will be conducted until data saturation has been reached, we estimate that we will conduct 12-15 interviews. The interviews will be analysed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease, with or without cognitive impairment
* People with Parkinson's living in their own home
* At least one fall in the preceding year, as reported by the person with Parkinson's or the caregiver
* Able to read a newspaper without severe difficulty, with or without glasses

OR

* An informal caregiver of a person with Parkinson's meeting the criteria for inclusion in the study

Exclusion Criteria:

* Diagnosis of a Parkinson's Plus syndrome
* People with Parkinson's living in a residential or nursing home
* No falls in the preceding year
* Non-fluent in verbal and written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of the guide | 3 months
  This will assessed through response to a questionnaire, with responses analysed through descriptive statistics
Feasibility and acceptability of the guide | 3 months
  A purposive sample of participants, selected through their responses to the questionnaire, will be invited to participate in semi-structured interviews. Interviews will explore the experiences and thoughts of the participants further and will be conducted until data saturation has been reached. Responses to the interview will be analysed through thematic analysis.

SECONDARY OUTCOMES:
Health related quality of life of people with Parkinson's as measured on PDQ8 | 3 months
  As measured on Parkinson's disease quality of life scale 8 (PDQ8)
Caregiver burden of their informal caregivers as measured on the Zarit Burden Interview scale short version | 3 months
  As measured on the Zarit Burden Interview scale short form

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No